CLINICAL TRIAL: NCT06777290
Title: Comparison of Whole-body MRI, Circulating DNA and PET-CT in Staging, Prognosis, and Treatment Response in Patients with Diffuse Large Cell B Lymphoma
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Lukas Lambert, prof. MD. Ph.D., Charles University, Czech Republic
Other Study IDs: 12/20 VFN IGP
Record Dates: First submitted 2024-12-06; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma, Diffuse Large B-Cell
Keywords: diagnostic performance; whole body MRI; PET/CT; ctDNA
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for circulating tumor DNA (ctDNA) analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DLBCL patients: Adult patients newly diagnosed with diffuse large cell B lymphoma

SUMMARY:
The aim of the study is to compare the diagnostic performance of whole-body MRI scan, positron emission tomography + CT, and circulating tumor DNA in patients with hematologic malignancy called diffuse large cell B lymphoma (DLBCL) in staging and restaging, and prognosis.

DETAILED DESCRIPTION:
Patients newly diagnosed with DLBCL or patients with relapsed DLBCL who consent to participate in this study will apart from standard staging and restaging examination with PET/CT undergo whole-body MRI (wbMRI). From blood samples, the level of circulating tumor DNA (ctDNA) fragments will be estimated. These procedures will be repeated during restaging after primary treatment. The diagnostic accuracy of wbMRI in initial staging and restaging will be compared with PET/CT as the gold standard. Circulating tumor DNA levels will be compared at baseline with staging from PET/CT. The change in levels of ctDNA will be compared with the treatement response assessed by PET/CT. All three methods will be used as prognostic indicators.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* performance status according to the Eastern Cooperative Oncology Group between 0 and 3
* satisfactory clinical condition to participate in this study
* adequate hematologic and renal functions
* no contraindications to MRI
* recent or planned PET/CT at the institution
* informed consent to participate.

Exclusion Criteria:

* history of indolent lymphoma
* anti-lymphoma treatment initiated before PET/CT or wbMRI
* central nervous system lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a Department of Hematology at a tertiary university hospital.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of whole-body MRI in staging of DLBCL | at baseline
  Comparison of diagnostic accuracy of whole-body MRI in staging of DLBCL in newly diagnosed adult patients before treatment compared to PET/CT as the gold standard

SECONDARY OUTCOMES:
Diagnostic value of MRI sequences | At baseline
  Rating of the diagnostic utility of MRI sequences used in whole body MRI in staging of DLBCL in newly diagnosed adult patients before treatment
Assessment of therapeutic response | after completion of first-line treatment, on average 6 months
  The assessment of therapeutic response by wbMRI after first-line treatment will be compared to that of PET/CT. Change in circulating tumor DNA will be correlated with therapeutic response assessed by PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Lambert, prof. M.D. Ph.D., Principal Investigator — Department of Radiology, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Czech Republic
Locations (1):
- Department of Radiology, General University Hospital in Prague, Prague, Czech Republic, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
The data will be available upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Lambert L, Burgetova A, Trneny M, Bircakova B, Molinsky J, Benesova K, Zogala D, Michalek P. The diagnostic performance of whole-body MRI in the staging of lymphomas in adult patients compared to PET/CT and enhanced reference standard-systematic review and meta-analysis. Quant Imaging Med Surg. 2022 Feb;12(2):1558-1570. doi: 10.21037/qims-21-649. PMID 35111648